CLINICAL TRIAL: NCT06028555
Title: International Active Surveillance Study: Native Estrogen Estetrol (E4) Safety Study
Acronym: INAS-NEES
Status: Recruiting | Type: Observational
Sponsor: Center for Epidemiology and Health Research, Germany (Other)
Collaborators: Estetra (Industry); Gedeon Richter Plc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ZEG2022_02
Record Dates: First submitted 2023-07-04; First posted 2023-09-08 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Contraception; Birth Control

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Estetrol/drospirenone (E4/DRSP): Users: Starters and re-starters
- Ethinyl estradiol/levonorgestrel (EE/LNG): Users: Starters and re-starters

SUMMARY:
Multinational, comparative, prospective, active surveillance study that follows two cohorts.

The primary objective of the study is to characterize and compare the risks of E4/Drospirenone (DRSP) with levonorgestrel-containing combined oral contraceptives (EE/LNG) in a study population that is representative of the actual users of these preparations. The main clinical outcome of interest is venous thromboembolism (VTE), specifically deep venous thrombosis (DVT) and pulmonary embolism (PE). Secondary objectives include measuring the occurrence of unintended pregnancy, assessing the risk of arterial thromboembolism (ATE), describing the drug utilization pattern, describing the baseline risk profile for VTE and ATE, and investigating outcomes associated with foetal exposure to E4/DRSP.

DETAILED DESCRIPTION:
Rationale and background:

The combined oral contraceptive (COC) containing estetrol (E4) and drospirenone (DRSP) (E4/DRSP) is a novel oral contraceptive containing a fixed dose of E4 (14.2 mg) and DRSP (3 mg). E4 is a natural oestrogen only produced during pregnancy by the foetal liver. When combined with the progestin DRSP, ovulation is inhibited. The E4/DRSP combination may have less impact on hepatic and haemostasis parameters in comparison to combinations of ethinyl estradiol (EE) and levonorgestrel (LNG) or EE and DRSP. Yet, it is unknown whether this regimen has an impact on the cardiovascular risk associated with the use of hormonal contraceptives.

Study design:

Multinational, comparative, prospective, active surveillance study that follows two cohorts. The cohorts consist of new users (starters and restarters ) of two different groups of hormonal contraceptives: E4/DRSP and EE/LNG. The study is taking a non-interventional approach to provide comprehensive information on these treatments in a routine clinical practice setting. Study participants will be enrolled via an international network of COC-prescribing health care professionals (HCPs) and then followed up for one to two years. All outcomes of interest will be captured by direct contact with the study participants. Reported outcomes of interest will be validated via attending physicians and relevant source documents. The classification of outcomes of interest into 'confirmed' and 'not confirmed' will be verified by blinded independent adjudication.

Population:

Approximately 101,000 study participants (50,500 E4/DRSP and 50,500 EE/LNG new users) will be recruited via a network of COC-prescribing health care professionals in Europe, the USA, and Brazil. All new users (starters and restarters) prescribed E4/DRSP or EE/LNG who are willing to participate may be eligible for enrolment in the study.

Data sources:

This is a field study that entails exposure to COCs and the occurrence of clinical outcomes of interest by completing questionnaires at baseline (study entry) and follow-up (at 6-, 12-, 18-, and 24-months post-baseline), in addition to potential confounding factors and potential effect modifiers. Medical confirmation of the occurrence of a clinical outcome of interest will be sought from the attending HCP and/or study participant (e.g., diagnostic report, discharge letter).

Study size:

The study is sufficiently powered to show non-inferiority of E4/DRSP compared to EE/LNG assuming that the VTE risk among E4/DRSP users is not higher than among EE/LNG users. For this purpose, a total of 101,000 women (50,500 E4/DRSP users and 50,500 EE/LNG users) will be recruited and followed up taking into account treatment adherence, treatment stopping/switching, and lost to follow-up (LTFU)/dropout.

Data analysis:

The final analyses will include both an "as-treated" (AT) and an "intention-to-treat" (ITT) analysis. All eligible women will be assigned to the ITT and AT population at baseline. Only women with follow-up information will be considered for longitudinal analysis. Women who never started their prescribed baseline medication will be considered in the ITT analysis but excluded from the AT analysis. Population characteristics, e.g., socio-economic factors, parameters of reproductive, contraceptive history, and medical history, will be summarized descriptively and used to estimate the probability of treatment differences. Inverse probability of treatment weighting combined with time-to-event analysis of VTE will be carried out based on the extended Cox model to calculate hazard ratios (HR) with 95% confidence intervals. The null hypothesis to be tested is HR of VTE ≥1.5 (i.e., the VTE HR for E4/DRSP vs. EE/LNG is higher than or equal to 1.5). The alternative hypothesis is HR of VTE <1.5.

ELIGIBILITY:
Inclusion Criteria:

New users of E4/DRSP New users of EE/LNG Germany: only recruitment of study participants who are prescribed the COC within on-label use

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 50,500 E4/ DRSP users and 50,500 EE/LNG new users, including adolescents (below the age of 18 years eligible based on local legislation) will be recruited via recruitment centres.
Sampling Method: Non-Probability Sample
Enrollment: 101000 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of Venous Thromboembolism (VTE) | Up to 24 months post baseline
  * Occurrence (or absence) of a new (non-recurrent) confirmed Deep Venous Thrombosis (DVT) of the lower extremities (International Classification of Diseases, 10th revision (ICD-10) codes: I80.1 and I80.2) and,
  * Occurrence (or absence) of a new (non-recurrent) confirmed Pulmonary Embolism (PE) (ICD-10 codes: I26.0 and I26.9)

SECONDARY OUTCOMES:
Incidence rate of all VTEs, including thromboses of the renal, mesenteric, portal, cerebral and retinal veins | Up to 24 months post baseline
  The occurrence (or absence) of a new (non-recurrent) confirmed VTE. A sensitivity analysis will be done for the ICD-10 code I80.3
Incidence rate of Arterial Thromboembolism (ATE), including acute myocardial infarction (AMI) and cerebrovascular accidents (CVA) | Up to 24 months post baseline
  The occurrence (or absence) of new (non-recurrent) confirmed ATE, AMI, and CVA: ICD-10 code I21; CVA: ICD-10 code: I24.9, G45.*, I61.*, I63.1, I63.2, I63.3, I63.4, I63.5, I63.8, I63.9
Incident rate of unintended pregnancy | Up to 24 months post baseline
  The occurrence of unintended pregnancy
Incident rate of neonatal malformations associated with foetal exposure to E4/DRSP and EE/LNG in E4/DRSP users and users of EE/LNG | Up to 24 months post baseline
  Occurrence of major congenital malformations, according to classification by the European network of population-based registries for the epidemiological surveillance of congenital anomalies (EUROCAT), as reported during follow-up among pregnancies observed
  * Stillbirth (defined as foetal death with a gestational age ≥20 weeks)
  * Neonatal death (defined as deaths occurring among live births during the first 28 completed days of life)
  * Spontaneous/elective abortion (defined as a loss of pregnancy at a gestational age <20 weeks)
  * Termination of pregnancy for foetal anomaly (TOPFA [where prenatal diagnosis was made of malformation in a live foetus and the pregnancy was then terminated])
  * Preterm delivery (defined as delivery strictly before 37 completed weeks of gestation)
  * Low birth weight (defined as a birth weight <2,500g)
  * Small for gestational age infants
Compare drug utilization pattern between users of both cohorts | Up to 24 months post baseline
  The time-varying exposure to COCs observed from study entry through the follow-up period, with dates and duration of each contraceptive prescription.

CONTACTS AND LOCATIONS:
Overall Officials: Klaas Heinemann, Dr., Principal Investigator — ZEG Berlin GmbH
Locations (1):
- Berlin Center for Epidemiology and Health Research, Berlin, State of Berlin, Germany